CLINICAL TRIAL: NCT03108937
Title: Effects of Serum From Patients Received Dexmedetomidine During General Anesthesia on Breast Cancer Cell Function in Vitro
Brief Title: Effects of Dexmedetomidine on Breast Cancer Cell Function in Vitro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DEX201703
Record Dates: First submitted 2017-04-06; First posted 2017-04-11 (Actual); Last update posted 2017-10-10 (Actual); Status verified 2017-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Experimental): Patients of dexmedetomidine group will receive a loading does of 1ug/kg dexmedetomidine since 15 mins before induction, and receive another 1ug/kg of dexmedetomidine at a rate of 0.5ug/kg/h for 2 continuous hours during surgery.
  Interventions: Drug: Dexmedetomidine
- saline (Placebo Comparator): Same amount of saline will be administrated.
  Interventions: Drug: saline

INTERVENTIONS:
Drug: Dexmedetomidine — Patients in the experimental group will receive Dexmedetomidine during surgery.
  Arms: Dexmedetomidine
Drug: saline — Patients in the control group will receive saline but not Dexmedetomidine during surgery.
  Arms: saline

SUMMARY:
Dexmedetomidine is widely used as an anaesthetic for general anesthesia during surgery. Previous studies in cells and animals show that dexmedetomidine may promote cancer growth. Using serum from breast cancer surgery patients randomized to receive dexmedetomidine or saline during surgery, we investigated the effects of dexmedetomidine on proliferation, migration and metastasis in MCF-7 breast cancer cells in vitro.

DETAILED DESCRIPTION:
Women diagnosed with breast cancer undergoing elective surgery under general anesthesia will be randomly allocated to dexmedetomidine group or control group. Patients from both groups will receive midazolam, propofol, fentanyl, remifentanil and CIS atracurium for total intravenous anesthesia. BIS value will be controlled between 40-60 during surgery. Patients of dexmedetomidine group will receive a loading does of 1ug/kg dexmedetomidine since 15 mins before induction, and receive another 1ug/kg of dexmedetomidine at a rate of 0.5ug/kg/h for 2 continuous hours during surgery. Patients of control group will receive same amount of normal saline. Serum will be collected from patients of both groups at before induction and 1h post-surgery. The MCF-7 breast cancer cell line will be treated with patient serum from both groups. The effects of dexmedetomidine on cellular proliferation, migration and metastasis will be measured.

ELIGIBILITY:
Inclusion Criteria:

* ASA grade I-III Age range of 18 to75 Patients diagnosed primary breast cancer(T2-3, N0-2, M0) Patients will have elective adenomammectomy

Exclusion Criteria:

* with history of breast operation Patients diagnosed carcinoma erysipelatodes Severe liver, renal, brain or lung disease with history of opioid addiction Patients diagnosed metastatic breast cancer

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2017-07-07 (Actual); Study Completion 2017-09-08 (Actual)

PRIMARY OUTCOMES:
cell proliferation | 24 hour post-surgery
  MCF-7 cells will be cultured with serum from patients of both groups for 24 hours and cell proliferation will be measured

SECONDARY OUTCOMES:
cell migration | 24 hour post-surgery
  MCF-7 cells will be cultured with serum from patients of both groups for 24 hours and cell migration will be measured
cell metastasis | 24 hour post-surgery
  MCF-7 cells will be cultured with serum from patients of both groups for 24 hours and cell metastasis will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Jie Tian, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu Y, Sun J, Wu T, Lu X, Du Y, Duan H, Yu W, Su D, Lu J, Tian J. Effects of serum from breast cancer surgery patients receiving perioperative dexmedetomidine on breast cancer cell malignancy: A prospective randomized controlled trial. Cancer Med. 2019 Dec;8(18):7603-7612. doi: 10.1002/cam4.2654. Epub 2019 Oct 30. PMID 31663690